CLINICAL TRIAL: NCT06806189
Title: Lipiodal Injection Technique for Free Flap Sparing Adjuvant Radiation Planning in Head and Neck Cancer
Brief Title: Lipiodal Injection Technique for Free Flap Sparing Adjuvant RT Planning in HNC
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Danielle MacNeil, Principal Investigator, Western University, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 126129
Record Dates: First submitted 2025-01-20; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Head and Neck Cancer
Keywords: Radiation planning; Head and neck cancer; Tumor delineation
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Intra-operative injection of lipiodal, a contrast agent (material injected to enhance x-ray and ct images) at the time of head and neck resection surgery to improve delineation of the interface between the removed mouth/throat cancer and the healthy tissue reconstructing the defect.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lipiodal injection (Experimental): Injection of contrast agent, Lipiodal, during surgical resection of head and neck cancer, for delineation of the interface between the removed mouth/throat cancer and the healthy tissue reconstructing the defect for radiation planning.
  Interventions: Drug: Lipiodal

INTERVENTIONS:
Drug: Lipiodal — Injection of lipiodal for delineation of interface between the removed mouth/throat cancer and the healthy tissue reconstructing the defect for radiation planning.

SUMMARY:
Patients with advanced mouth/throat cancers require surgery to remove the cancer followed by reconstruction with transplanted skin/muscle/bone from another location in their body to restore function. This is called a free-flap (skin/muscle/bone used from another part of the body to reconstruct the cancer site). Post-operative radiation therapy is often recommended to reduce the risk of cancer coming back. Unfortunately, radiation can exacerbate issues with swallowing and speech and lead to other complications. To date, there has been no mechanism to allow sparing of the healthy tissue from radiation while ensuring delivery to all at-risk areas.

This is a proof-of-principle study that injects a safe contrast agent (material injected to enhance x-ray and ct images) at the time of surgery to improve delineation of the interface between the removed mouth/throat cancer and the healthy tissue reconstructing the defect. In doing so, the investigators hope to demonstrate the potential to spare post-operative radiation to the healthy reconstructive tissue and improve patient function.

The investigators propose using Lipiodal, a poppyseed oil-extract that has been in safe clinical use for > 100-years, in 10 patients. There will be no change to the way in which patients are treated for their mouth/throat cancer or in the way radiation is delivered. The investigators will assess the feasibility and safety of injecting Lipiodal at the time of surgery and visualization on post-operative CT scans. This has been shown to be both safe and feasible in patients with other cancers, such as bladder cancer, however patients will be closely monitored for any side effects. Patients will provide informed consents and be able to withdraw at any time.

DETAILED DESCRIPTION:
Lipiodal is approved and indicated for subcutaneous injection in children and adults for the purposes of lymphatic mapping.12 Free flap reconstruction in the head and neck typically uses fasciocutaneous flap comprising skin, dermis, subcutaneous tissue and deep fascia. Composite reconstructions can also include vascularised muscle and bone. Bone margins are well defined on pre- and post-operative imaging. However, it is the soft tissue muco-cutaneous margins in the oral cavity and pharynx in particular that are less reliable on post operative imaging due to effects of post-operative edema and gravity/positional dependence. Thus, injecting a liquid fiducial marker such as Lipiodal to the margins of the free flap in the dermal/subcutaneous plane will be of maximal benefit in delineating margins of healthy flap tissue and tumour bed for the purposes of post-operative radiation planning. This type of injection to the dermal/subcutaneous tissue is currently routinely performed in interventional radiology at London Health Sciences Centre at Victoria Hospital for lymphography and meets with approved clinical indications for use in Canada and at our institution.

Ten patients with locally advanced (T2-T4) oral cavity squamous cell carcinoma undergoing primary surgical resection with free flap reconstruction and adjuvant radiation therapy will be recruited for the study and treated with standard of care surgery and adjuvant treatment as per the London Regional Cancer Program Head and Neck Tumour Board recommendations at Victoria Hospital. Patients with previously treated locally advanced head and neck malignancy (either with surgery and/or radiotherapy) will be excluded from the study. Patients not requiring free flap reconstruction will be excluded from the study.

Patients will be injected with Lipiodal at the time of resection of their head and neck tumours. Injections will be delivered using a 22G needle on a 10ml syringe. Each injection will be 0.5ml aliquot delivered trans epidermal to the subcutaneous margin of the free flap, 2-3mm within the free margin. This will provide constancy in tissue type being injected and allow visualisation of an epidermal wheal as confirmation of successful injection. This volume will allow up to 20 injections to be equally spaced circumferentially around the free flap thus defining the interface with the tumour bed.

Patients will be followed closely post-operatively as an inpatient for 7-14 days as per standard of care with at least twice daily visual reviews of the flap, assessing perfusion, inflammatory change (such as dermatitis or lipogranuloma) and healing progress at the flap inset margin. Early post-operative CT scan will be performed at day 5 post-op as per standard of care, which will opportunistically allow assessment of Lipiodal delivery to the tumour-bed/free-flap interface and also ensure no local complication. Upon discharge, patients will be followed closely with reviews at 1-, 4-, and 8-weeks post-operatively as per standard of care. Patients will receive a post-operative planning CT scan under the supervision of the treating radiation oncologist as per standard of care at 6-8 weeks post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years and older) seen at the head and neck clinic at London Health Sciences Centre (LHSC)
* Locally advanced T2-4N0-3M0 mucosal or cutaneous squamous cell carcinoma involving the oral cavity requiring composite resection and free flap reconstruction

Exclusion Criteria:

* Previous treated locally advanced head and neck cancer with surgery and/or radiation
* History of hypersensitivity or adverse reaction to Lipiodal or any iodinated radiocontrast
* Severe bronchial asthma
* Severe renal dysfunction
* Hyperthyroidism
* Pregnant
* Breastfeeding
* Clinically apparent cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Success of intra-operative injection | Intra-operative
  Successful or unsuccessful injection of Lipiodal
Success of visualisation on immediate post-operative and adjuvant radiation planning CT scans | Day 5 post-op CT and 6-8 week post-operative radiation planning CT scan
  Success of visualisation of tumour bed-free flap interface

SECONDARY OUTCOMES:
Complications of injection to the flap tissue | Intra-operatively, immediately post-operatively, through study completion, an average of 6 months
  dermatitis, lymphangitis, disproportionate oedema, lipogranuloma, delayed healing, dehiscence
Safety outcomes | Immediately post-operatively, through study completion, an average of 6 months
  Any adverse events graded per CTCAE criteria, any evidence allergic/anaphylactoid reaction

CONTACTS AND LOCATIONS:
Overall Officials: Danielle MacNeil, MD, Principal Investigator — Department of Otolaryngology-Head & Neck Surgery, Western University Canada
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Data will be made available upon request